CLINICAL TRIAL: NCT05536141
Title: A Phase 1, Open-label, Dose Escalation and Dose Expansion Study, to Investigate the Safety, Tolerability, and Pharmacokinetic Profile of AB521 Monotherapy and Combination Therapies in Participants With Clear Cell Renal Cell Carcinoma and Other Solid Tumors
Brief Title: A Phase 1 Study of AB521 Monotherapy and Combination Therapies in Renal Cell Carcinoma and Other Solid Tumors
Acronym: ARC-20
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Arcus Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ARC-20; 2024-519142-70-00 (EU CTIS Number)
Record Dates: First submitted 2022-09-07; First posted 2022-09-10 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-04

CONDITIONS: Clear Cell Renal Cell Carcinoma; Solid Tumors
Keywords: Clear Cell Renal Cell Carcinoma; Solid Tumor Malignancies; AB521; Casdatifan; Kidney Cancer; Zimberelimab; AB122
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms | interventions — cabozantinib; zimberelimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (13):
- Dose Escalation Cohort 1 (Experimental): Participants will receive casdatifan orally once daily
  Interventions: Drug: casdatifan
- Dose Escalation Cohort 2 (Experimental): Participants will receive casdatifan orally once daily
  Interventions: Drug: casdatifan
- Dose Escalation Cohort 3 (Experimental): Participants will receive casdatifan orally twice daily
  Interventions: Drug: casdatifan
- Dose Escalation Cohort 4 (Experimental): Participants will receive casdatifan orally once daily
  Interventions: Drug: casdatifan
- Dose Escalation Cohort 5 (Experimental): Participants will receive casdatifan orally once daily
  Interventions: Drug: casdatifan
- Dose Expansion Cohort 1 (Experimental): Participants will receive casdatifan orally
  Interventions: Drug: casdatifan
- Dose Expansion Cohort 2 (Experimental): Participants will receive casdatifan orally
  Interventions: Drug: casdatifan
- Dose Expansion Cohort 3 (Experimental): Participants will receive casdatifan orally
  Interventions: Drug: casdatifan
- Dose Expansion Cohort 4 (Experimental): Participants will receive casdatifan orally with with cabozantinib orally
  Interventions: Drug: casdatifan; Drug: Cabozantinib
- Dose Expansion Cohort 5 (Experimental): Participants will receive casdatifan orally
  Interventions: Drug: casdatifan
- Dose Expansion Cohort 6 (Experimental): Participants will receive casdatifan orally
  Interventions: Drug: casdatifan
- Dose Expansion Cohort 7 (Experimental): Participants will receive casdatifan orally with zimberelimab infusion
  Interventions: Drug: casdatifan; Drug: Zimberelimab
- Dose Expansion Cohort 8 (Experimental): Participants will receive casdatifan orally
  Interventions: Drug: casdatifan

INTERVENTIONS:
Drug: casdatifan — Administered as specified in the treatment arm
  Other Names: AB521
Drug: Cabozantinib — Administered as specified in the treatment arm
  Arms: Dose Expansion Cohort 4
Drug: Zimberelimab — Administered as specified in the treatment arm
  Other Names: AB122
  Arms: Dose Expansion Cohort 7

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of:

* casdatifan when taken alone in participants with advanced solid tumor malignancies and clear cell renal cell carcinoma (ccRCC) during the dose escalation stage; and
* casdatifan monotherapy and casdatifan in combination with cabozantinib or zimberelimab in participants with ccRCC in the dose expansion stage

ELIGIBILITY:
Key Inclusion Criteria:

* Must have at least one measurable lesion per RECIST guidance
* Eastern Cooperative Oncology Group (ECOG) performance status score of ≤ 1
* Disease-specific criteria for dose escalation:

  * Participants may have any pathologically confirmed solid tumor type where no other treatment options are available
  * Creatinine clearance ≥ 40 mL/min

Disease-specific criteria for dose-expansion:

* Histologically confirmed ccRCC
* Creatinine clearance ≥ 40 mL/min

Key Exclusion Criteria:

* Use of any live vaccines against infectious diseases (eg, influenza, varicella) within 4 weeks (28 days) of initiation of investigational product
* Has any other clinically significant cardiac, respiratory, or other medical or psychiatric condition that might interfere with a participant's participation in the clinical study or make the administration of investigational product hazardous
* History of trauma or major surgery within 28 days prior to the first dose of investigational product
* For all expansion cohorts: prior treatment with an hypoxia inducible factor (HIF)-2α inhibitor. For the casdatifan + cabozantinib combination cohort, any prior treatment with cabozantinib
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Estimated)
Dates: Start 2022-10-26 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Number of participants with dose limiting toxicities (DLTs) | Up to 4 months
Number of participants with adverse events (AEs) | Up to 4 months

SECONDARY OUTCOMES:
Objective Response Rate as measured by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 | Up to 4 months
Plasma concentration of casdatifan | Up to 4 months
Area under the plasma concentration time curve (AUC) of casdatifan | Up to 4 months
Maximum Observed Plasma Concentration (Cmax) of casdatifan | Up to 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Arcus Biosciences
Locations (29):
- United States (20):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California at San Diego, San Diego, California
  - UCLA, Santa Monica, California
  - University of Miami, Miami, Florida
  - Emory University, Atlanta, Georgia
  - University of Louisville Brown Cancer Center, Louisville, Kentucky
  - Oschner Health, New Orleans, Louisiana
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Center, Detroit, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Nebraska Cancer Specialists - Oncology Hematology West PC, Omaha, Nebraska
  - Tisch Cancer Institute, Icahn Mount Sinai Hospital, New York, New York
  - Memorial Sloan Kettering, New York, New York
  - University Hospitals Cleveland Clinical, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Sarah Cannon, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - South Texas Accelerated Research Therapeutics, LLC, San Antonio, Texas
- Australia (4):
  - Chris O'Brien Lifehouse, Camperdown
  - Box Hill Hospital, Melbourne
  - Ashford Cancer Centre Research/ICON, Sydney
  - Macquarie University Hospital, Sydney
- South Korea (4):
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Bundang Hospital, Seoul
  - Severance Hospital, Seoul
- Vall d'Hebron Institute of Oncology (VHIO), Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Arcus will provide access to individual de-identified participant data and related study documents [e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)] upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions.
  For more information, please visit our website.
Supporting Information: Study Protocol, SAP, CSR
URL: https://trials.arcusbio.com/our-transparency-policy

REFERENCES:
- See also: ARC-20 - Public website — https://trials.arcusbio.com/study/?id=ARC-20